CLINICAL TRIAL: NCT06461715
Title: Left Bundle Branch Area Pacing Study Designing the 3D Hybrid Guidance System for Implantation of Cardiac Devices
Brief Title: Left Bundle Branch Area Pacing 3D Guidance System
Status: Not yet recruiting | Type: Observational
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 333704
Record Dates: First submitted 2024-06-05; First posted 2024-06-17 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Left Bundle Branch Pacing; Heart Failure; Bradycardia
Keywords: Left bundle branch pacing; Pacemaker; Artificial intelligence; Conduction system pacing
MeSH Terms: conditions — Heart Failure; Bradycardia | interventions — Machine Learning

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Left bundle branch pacing group: Patients who underwent left bundle branch pacing
  Interventions: Other: Machine learning with artificial intelligence software program

INTERVENTIONS:
Other: Machine learning with artificial intelligence software program — This is a retrospective observational study using cardiac MRI, cardiac CT and x-ray fluoroscopy images to develop a 3D hybrid guidance system with the use of deep learning methods.

SUMMARY:
The investigator's project proposes the development of a 3D hybrid guidance system which has the aim of avoidance of scar and septal perforation through targeted lead deployment via a personalised septal real time image overlay onto x-ray fluoroscopy imaging during left bundle branch pacing. The investigators hypothesise that the use of cardiac anatomy and myocardial scar distribution derived from cardiac magnetic resonance imaging (MRI) as well as 3D position of the pacing lead, may improve LBBAP lead deployment success and improve clinical outcomes by guiding the physician towards optimal lead positioning.

DETAILED DESCRIPTION:
The study will use anonymised imaging data from the TACTIC-CRT (IRAS 250715) , Cardiac CT to guide Cardiac Resynchronisation Therapy (CRT) implantation (IRAS 150161) study (IRAS 150161) and anonymous cardiac MRI, CT and fluoroscopy imaging data from patients who underwent LBBA pacing to develop a 3D hybrid guidance system using machine learning methods. The developed 3D hybrid guidance system will be tested on anonymised retrospectively collected x-ray fluoroscopy images from patients who underwent LBBAP and had a cardiac MRI. The 3D hybrid guidance system will collect data from the retrospective anonymised X-ray fluoroscopic images, detect the pacing lead and reconstruct the 3D position of the pacing lead and test the accuracy of the 3D hybrid guidance system.

ELIGIBILITY:
Inclusion Criteria:

* All patients who took part in the TACTIC-CRT (IRAS 250715) and Cardiac CT to guide Cardiac Resynchronisation Therapy (CRT) implantation (IRAS 150161) study.
* All patients who received a LBBA pacing device from the GSTT/RBH/ICH database in the last 10 years (from 01/01/2014) and had a cardiac MRI for assessment of scar.
* All patients who are >18 years old.
* Male and Female

Exclusion Criteria:

* All patients <18 years old
* Patients with congenital heart disease
* Patients who did not have a cardiac MRI before receiving a LBBA pacing device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Anonymised images from patients who took part in the TACTIC-CRT (IRAS 250715) and Cardiac CT to guide Cardiac Resynchronisation Therapy (CRT) implantation (IRAS 150161) or who received left bundle branch pacing and had a cardiac MRI
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Detection of the position of the left bundle branch area on x-ray fluoroscopy | 12 months
  The accuracy of left bundle branch area detection will be measured as intersection-over-union (IoU) with the use of a convolutional neural network

CONTACTS AND LOCATIONS:
Locations (1):
- Imperial College Nhs Healthcare Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No